CLINICAL TRIAL: NCT03577132
Title: The Efficacy of Neoadjuvant Atezolizumab Treatment in Patients With Advanced Urothelial Bladder Cancer According to the BASQ Classification
Brief Title: The Efficacy of Neoadjuvant Atezolizumab Treatment in Patients With Advanced Urothelial Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ja Hyeon Ku, Professor, MD., PHD., Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SeoulNUHUro_Atezolizumab
Record Dates: First submitted 2018-06-24; First posted 2018-07-05 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Urothelial Carcinoma
Keywords: neoadjuvant chemotherapy; atezolizumab
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luminal type (Experimental): Luminal type in previous transurethral resection of bladder tumor pathology. Luminal type in Immunohistochemistry (KRT5/6-KRT14-FOXA1+GATA3+)
  Interventions: Drug: Neoadjuvant atezolizumab
- Basal typr (Experimental): Basal type in previous transurethral resection of bladder tumor pathology. Basal type in Immunohistochemistry (KRT5/6+KRT14+FOXA1-GATA3-)
  Interventions: Drug: Neoadjuvant atezolizumab

INTERVENTIONS:
Drug: Neoadjuvant atezolizumab — Atezolimumab
  * At a fixed dose of 1200 mg as a 60-minute intravenous infusion (1st), then as a 30-minute intravenous infusion (2nd and 3rd)
  * Every 3 weeks, for a total of 3 cycles prior to radical cystectomy

SUMMARY:
Recently, promising evidences that blocking PD-1 and PD-L1 is an efficacious way to treat advanced stage bladder cancer patients. Atezolimumab is the first PD-L1 inhibitor approved by US FDA for advanced UBC in June 2014. These novel agents will become the standard therapy for unhopeful UBC patients who fail to respond to cisplatin-based chemotherapy and finally, the first-line treatment would be changed from cisplatin-based chemotherapy to immune check point inhibitors for advanced UBC, particularly neoadjuvant setting.

Additionally, along with enormous analysis of genomic landscape of bladder cancer, a consensus was reached regarding the existence of a group of Basal-Squamous-like tumors - designated BASQ - characterized the high expression of KRT5/6 and KRT14 and low/undetectable expression of FOXA1 and GATA3. This novel molecular classification can improve the identification of optimal patient population for different treatment modalities. Specifically, luminal type and basal type may have different treatment response and prognosis after initial definitive treatment, such as neoadjuvant treatments.

However, there is no evidence for this topic, particularly the clinical efficacy of neoadjuvant PD-L1 inhibitors according to the BASQ classification in patients with advanced urothelial bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Histologically confirmed muscle-invasive urothelial carcinoma
* Patients undergoing radical cystectomy
* Advanced status requiring neoadjuvant systemic therapy
* ECOG performance status score of 0 or 1
* Adequate organ and hematologic functions
* Available IHC data for the BASQ classification

Exclusion Criteria:

* Non-urothelial carcinoma histology
* Active autoimmune disease or inflammatory bowel disease
* Prior severe or persistent immune-related adverse events
* Previous exposure to anti-PD-1 or anti-PD-L1 therapy
* Requirement for 10 mg/d of prednisone or equivalent
* Inadequate liver, kidney function and hematologic dysfunction
* Inoperable case, such as untreated CNS metastases
* No available archival tumor tissue for evaluating the BASQ classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
objective pathological responses (pT0 change) | 4weeks
  Final pathology of bladder after operation (radical cystectomy)

SECONDARY OUTCOMES:
progression-free survival at 1yr | 1year
  progression-free survival at 1yr

CONTACTS AND LOCATIONS:
Overall Officials: Ja Hyeon Ku, M.D.,PH.D, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grossman HB, Natale RB, Tangen CM, Speights VO, Vogelzang NJ, Trump DL, deVere White RW, Sarosdy MF, Wood DP Jr, Raghavan D, Crawford ED. Neoadjuvant chemotherapy plus cystectomy compared with cystectomy alone for locally advanced bladder cancer. N Engl J Med. 2003 Aug 28;349(9):859-66. doi: 10.1056/NEJMoa022148. PMID 12944571
- [Background] von der Maase H, Sengelov L, Roberts JT, Ricci S, Dogliotti L, Oliver T, Moore MJ, Zimmermann A, Arning M. Long-term survival results of a randomized trial comparing gemcitabine plus cisplatin, with methotrexate, vinblastine, doxorubicin, plus cisplatin in patients with bladder cancer. J Clin Oncol. 2005 Jul 20;23(21):4602-8. doi: 10.1200/JCO.2005.07.757. PMID 16034041
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of urothelial bladder carcinoma. Nature. 2014 Mar 20;507(7492):315-22. doi: 10.1038/nature12965. Epub 2014 Jan 29. PMID 24476821
- [Background] Choi W, Czerniak B, Ochoa A, Su X, Siefker-Radtke A, Dinney C, McConkey DJ. Intrinsic basal and luminal subtypes of muscle-invasive bladder cancer. Nat Rev Urol. 2014 Jul;11(7):400-10. doi: 10.1038/nrurol.2014.129. Epub 2014 Jun 24. PMID 24960601
- [Background] Balar AV, Galsky MD, Rosenberg JE, Powles T, Petrylak DP, Bellmunt J, Loriot Y, Necchi A, Hoffman-Censits J, Perez-Gracia JL, Dawson NA, van der Heijden MS, Dreicer R, Srinivas S, Retz MM, Joseph RW, Drakaki A, Vaishampayan UN, Sridhar SS, Quinn DI, Duran I, Shaffer DR, Eigl BJ, Grivas PD, Yu EY, Li S, Kadel EE 3rd, Boyd Z, Bourgon R, Hegde PS, Mariathasan S, Thastrom A, Abidoye OO, Fine GD, Bajorin DF; IMvigor210 Study Group. Atezolizumab as first-line treatment in cisplatin-ineligible patients with locally advanced and metastatic urothelial carcinoma: a single-arm, multicentre, phase 2 trial. Lancet. 2017 Jan 7;389(10064):67-76. doi: 10.1016/S0140-6736(16)32455-2. Epub 2016 Dec 8. PMID 27939400
- [Derived] Yuk HD, Jeong CW, Kwak C, Kim H, Moon KC, Ku JH. Efficacy of neoadjuvant atezolizumab treatment in patients with advanced urothelial bladder cancer according to the BASQ classification: a study protocol for an open-label, two-cohort, phase II trial. BMJ Open. 2020 Oct 15;10(10):e035530. doi: 10.1136/bmjopen-2019-035530. PMID 33060077